CLINICAL TRIAL: NCT07348731
Title: Comparison of the Effects of Foot Bath, ShotBlocker®, and Buzzy® on Neonatal Vital Signs During Heel Lance
Brief Title: Non-Pharmacological Methods in Heel Lance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Sermin Dinc, Assistant Professor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-22686390-050.99-84286
Record Dates: First submitted 2025-12-06; First posted 2026-01-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heel Lance Procedures
Keywords: Foot Bath; Buzzy; Shotblocker; heel lance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buzzy (Experimental): Vibration Application with Buzzy® Before Heel Lance
  Interventions: Behavioral: Foot bath
- Shotblocker (Experimental): After the information form is completed with the parent, the video recording will be initiated. The infant's vital signs will be monitored and recorded using a pulse probe, after which the ShotBlocker® will be placed on the procedure site. Following the heel lance performed with the ShotBlocker®, the time to bleeding cessation and the infant's crying duration will be recorded.
  Interventions: Behavioral: Foot bath

INTERVENTIONS:
Behavioral: Foot bath — The infant's foot designated for blood sampling will be immersed up to the mid-calf level in water adjusted to 37-38°C, using a thermometer for confirmation, and kept there for 5 minutes.
  The heel lance procedure will then be performed by the nurse working in the clinic, following the standard clinical routine.
  The video recording will be stopped once bleeding has ceased at the end of the procedure.
  The video recordings obtained before, during, and after the procedure will be reviewed, and the infant's pain scores will be assessed by two independent experts.

SUMMARY:
This randomized controlled study was designed to compare the effects of Warm Foot Bath, ShotBlocker®, and Buzzy®-applied prior to heel lance-on the vital signs of newborns. Heel lance is one of the most frequently performed invasive procedures during the neonatal period, and the pain and stress experienced during the procedure may lead to alterations in vital parameters such as heart rate, respiratory rate, and oxygen saturation. Therefore, identifying non-pharmacological, safe, and feasible pain management methods is essential for enhancing the quality of nursing care.

Data will be collected at three time points: before, during, and after the procedure, and changes in heart rate, respiratory rate, and SpO₂ will be recorded. With parental consent, the procedure will be video-recorded before, during, and after heel lance; the recordings will be anonymized and shared with experts for pain assessment. Additionally, the infant's crying duration and time to bleeding cessation will also be evaluated.

DETAILED DESCRIPTION:
This study was designed to investigate the effects of three different non-pharmacological interventions applied prior to heel lance on the vital parameters and pain levels of newborns. The study population consists of term newborns who meet the inclusion criteria, and the sample includes newborns who present with their parents to a state hospital for heel lance and meet these criteria. Following ethical approval, data will be collected between November 2025 and November 2026. Data collection will be carried out by Özlem Kum, a graduate student actively working in the relevant clinic and responsible for performing the procedures.

Pain will be assessed using the Neonatal Infant Pain Scale (NIPS), which evaluates procedural pain in both preterm and term newborns. The scale includes five behavioral indicators (facial expression, leg movement, arm movement, crying, and state of arousal) and one physiological indicator (respiratory pattern), with total scores ranging from 0 to 7. A 16-item Information Form containing maternal and neonatal characteristics will also be used. Statistical analyses will be performed using SPSS version 26, including frequency, percentage, mean, standard deviation, t-test, ANOVA, and Pearson correlation analyses.

Heel lance is one of the most frequently performed invasive procedures in the neonatal period. The pain and stress experienced during this procedure may lead to changes in vital parameters such as heart rate, respiratory rate, and oxygen saturation. Therefore, identifying non-pharmacological, safe, and feasible pain management strategies is essential for improving the quality of nursing care.

Non-pharmacological methods such as warm foot bath, ShotBlocker®, and the Buzzy® device are commonly used to reduce procedural pain through different mechanisms, including increased peripheral circulation, mechanical stimulation, vibration, and cold application. However, studies comparing the effects of these methods on newborns' heart rate, respiratory rate, oxygen saturation, and pain levels are limited.

This study will be conducted with approximately 90 clinically stable term newborns (37-42 weeks of gestation) in the Neonatal Unit of Kocaeli City Hospital. Data will be collected at three time points-before, during, and after the procedure-and changes in heart rate, respiratory rate, and oxygen saturation will be recorded. With parental consent, the procedure will be video-recorded at all stages, and anonymized recordings will be shared with experts for pain assessment.

The findings of this study are expected to contribute to the identification of effective non-pharmacological methods that can be used during painful procedures such as heel lance and to support the development of evidence-based practices in neonatal nursing.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with a gestational age of ≥37 weeks
* Newborns in the neonatal period (0-28 days)
* Stable vital signs
* Obtained informed consent from the parents
* No use of analgesics or sedatives within the 24 hours before the procedure
* Absence of any respiratory problems
* First-time heel lance procedure
* No condition that would interfere with pain assessment

Exclusion Criteria:

* Preterm or low birth weight infants (< 2500 g)
* Infants with congenital anomalies or requiring respiratory support
* Infants receiving sedative or analgesic treatment

Ages: 4 Days to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale | 0 minutes (T0)
  Min. 0-Max. 7 points (0-2 = mild to no pain, 3-4 = mild to moderate pain, >4 = severe pain) moderate pain, >4 = severe pain)
Neonatal Infant Pain Scale | 5th minutes 1st (T1)
  Min. 0-Max. 7 points (0-2 = mild to no pain, 3-4 = mild to moderate pain, >4 = severe pain)
Neonatal Infant Pain Scale | 10th minutes (T2)
  Min. 0-Max. 7 points (0-2 = mild to no pain, 3-4 = mild to moderate pain, >4 = severe pain)
Heart Rate | 0 min (T0)
  beats/min.
Heart Rate | 5th min 1st (T1)
  beats/min.
Heart Rate | 10th minutes (T2)
  beats/min.
Respiratory rate | 0 min (T0)
  respiration/minute
Respiratory rate | 5th min 1st (T1)
  respiration/minute
Respiratory rate | 10th minutes (T2)
  respiration/minute
Saturation level | 0 min (T0)
  %100
Saturation level | 5th min 1st (T1)
  %100
Saturation level | 10th minutes (T2)
  %100

SECONDARY OUTCOMES:
The infant's crying duration | From start to end of the procedure
  minutes

OTHER OUTCOMES:
Duration of the procedure | From start to end of the procedure
  minutes

CONTACTS AND LOCATIONS:
Overall Officials: sermin dinç, Dr., Principal Investigator — Atlas University
Locations (1):
- Atlas University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effect of the ShotBlocker® and breastfeeding on pain and comfort level during heel lance procedure in newborns: randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/40716331